CLINICAL TRIAL: NCT00330603
Title: Serial Exhaled Breath pH Monitoring
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Virginia (Other)
Responsible Party: John Hunt, MD, University of Virginia, Pediatrics
Other Study IDs: 12302
Record Dates: First submitted 2006-05-26; First posted 2006-05-29 (Estimated); Last update posted 2011-03-08 (Estimated); Status verified 2011-03

CONDITIONS: Gastroesophageal Reflux
Keywords: Cough; Gastroesophageal Reflux
MeSH Terms: conditions — Gastroesophageal Reflux; Cough

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

INTERVENTIONS:
Procedure: Serial exhaled breath collections — collect breath for 5 minutes on 8 occasions

SUMMARY:
This study will seek to determine the amount of acids a person with a chronic cough that is suspected to be related to acid reflux breathes out after coughing. The study will also seek to determine if this measurement can predict the best treatment for the cough.

Subjects with a chronic cough which is suspected to be related to acid reflux for which their doctor has prescribed a proton pump inhibitor medication will be enrolled in this study.

DETAILED DESCRIPTION:
Acid reflux has been considered to be a key contributor to cough, particularly in patients with obstructive lung diseases. However, diagnosis has relied upon either responsiveness to high dose twice daily administration of proton pump inhibitor therapy or by 24 hour esophageal pH probes. This study is designed to provide information for the development of a clinically useful diagnostic (exhaled breath condensate pH) to identify the contribution of acid reflux to cough.

Exhaled breath condensate (EBC) pH has been well documented to reflect airway acidification. Acid reflux to the level of the hypopharynx, which is a key common trigger of acid reflux induced cough, acidifies the airway sufficiently to be identified with EBC pH assays. The association of low EBC pH with an immediately preceding cough strongly suggests an association of the cough with an airway acid event, and even if the acidity is not prolonged, acid reflux becomes highly suspect.

This study will examine the ability of EBC pH measurements to prognose the likelihood of a positive response to acid blockade with proton pump inhibitor therapy in subjects with chronic cough.

ELIGIBILITY:
Inclusion Criteria:

* Outpatient
* 5 years of age and older
* Cough lasting a minimum of 3 weeks
* Has been prescribed a proton pump inhibitor as a single therapeutic and diagnostic effort to control the cough

Exclusion Criteria:

* Inability to perform serial exhaled breath condensate collections at home
* Unwillingness to initiate proton pump inhibitor therapy as prescribed by physician
* Other changes planned in therapy, such as initiating or discontinuing cough suppressant therapy, initiating or augmenting antibiotic therapy, initiating or augmenting anti-inflammatory therapy
* Previous treatment of respiratory symptoms with proton pump inhibitor therapy
* Current treatment with angiotensin converting enzyme inhibitor medication or H2 antagonists
* Regular exposure to an environmental irritant

Min Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients with chronic cough for whom their doctor is planning to begin an empiric trial of proton pump inhibitor as a diagnostic trial of therapy.
Sampling Method: Non-Probability Sample
Enrollment: 99 (Estimated)
Dates: Start 2006-04; Primary Completion 2011-12 (Estimated); Study Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
pH of cough samples | 1 month
change in Leicester Cough Questionnaire (LCQ) total score | 1 month

SECONDARY OUTCOMES:
proton pump inhibitor dosing | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: John Hunt, MD, Principal Investigator — University of Virginia
Locations (1):
- University of Virginia, Charlottesville, Virginia, United States